CLINICAL TRIAL: NCT06779006
Title: Effectiveness of Internet-Based Self-Help ACT With Behavioral Activation in Improving Alcohol Use Abstinence Among Ethnic Minority Young Adults With Alcohol Use Disorder in Hong Kong, 2024: A Pilot Randomized Controlled Trial
Brief Title: Effectiveness of Internet-Based Self-Help ACT With Behavioral Activation in Improving Alcohol Use Abstinence Among Ethnic Minority Young Adults With Alcohol Use Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Eva Ho, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ACT-BA_AUD
Record Dates: First submitted 2024-08-28; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder
Keywords: Acceptance and commitment therapy; Behavioral activation; Ethnic minority young adults; Alcohol abuse; Alcohol use disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The intervention group will receive online-based integrated ACT with BA therapy. The protocol of this therapy is adapted from the ACT manual, self-help protocols for mental health problems, and behavioral activation treatment for substance use and depression.
  Interventions: Behavioral: Self-help acceptance and commitment therapy with behavioral activation
- Control Arm (No Intervention): The control group will be assigned to receive Treatment as Usual (TAU).

INTERVENTIONS:
Behavioral: Self-help acceptance and commitment therapy with behavioral activation — Internet-based self-help acceptance and commitment therapy with behavioral activation
  Arms: Intervention Arm

SUMMARY:
The goal of this clinical trial is to examine the preliminary effectiveness and feasibility of internet-based self-help acceptance and commitment therapy with behavioral activation for ethnic minority young adults with alcohol use disorder. The main questions it aims to answer are:

* Is the internet-based self-help acceptance and commitment therapy with Behavioral activation (self-help iACT-BA) feasible and acceptable for ethnic minority young adults with AUD?
* Does the self-help iACT-BA promote greater abstinence from alcohol use compared to treatment as usual (TAU) in ethnic minority young adults diagnosed with AUD? Researchers will compare self-help iACT-BA to treatment as usual (TAU) to see if self-help iACT-BA works to treat alcohol use disorder in ethnic minority young adults.

Participants will:

* Received a self-help iACT-BA module every week for 6 weeks. or a placebo every day for 4 months
* Access the module every week, read the material, practice, and complete home assignments.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong ethnic minority young adults
* They have to read, write, and speak English
* Their age will range from 18 to 25
* They will be voluntary to participate
* Participants should have smartphones or other electronic devices to access the internet
* They must have AUD based on DSM-5 criteria.

Exclusion Criteria:

* Currently having psychiatric problems, other mental health problems, being actively involved in suicidal attempts, or immediate care
* Having a plan to go out of Hong Kong during intervention implementation
* Having no access to the internet, smart telephone, or other electronic devices
* Have participated in another psychosocial or pharmacological intervention for AUD.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-03-28 (Estimated); Study Completion 2025-04-28 (Estimated)

PRIMARY OUTCOMES:
Screening rate | 3 months
  calculated as the number of Hong Kong ethnic minority young adults screened by the research assistant divided by the number of Hong Kong ethnic minority young adults available for screening during the recruitment period.
Eligibility rate | 3 months
  Calculated as the number of eligible ethnic minority young adults divided by the number of screened ethnic minority young adults.
Consent rate | 3 months
  calculated as the number of eligible ethnic minority young adults who join the study divided by the number of eligible ethnic minority young adults.
Randomization rate | 2 weeks
  calculated as the number of ethnic minority young adults who are randomized into the experimental and control groups, divided by the number of eligible ethnic minority young adults who consent to join the study
Attendance rate | 6 weeks
  calculated as the number of subjects in the experimental group who complete the intervention divided by the number of subjects randomized into the experimental group.
Adherence rate | 6 weeks
  calculated as the number of subjects in the experimental group who practice the ACT skills gained in the intervention divided by the number of subjects randomized into the experimental group
Retention rate | 6 weeks
  calculated the number of subjects who remain in the study, divided by the number of subjects who are randomized
Completion rate | 6 weeks
  calculated as the number of subjects who answer the questionnaires divided by the number of questionnaires distributed
Missing data | 6 weeks
  percentage of missing in the dataset. Unknown or blank values will be regarded
Adverse events | 6 weeks
  unfavorable and unintended events that are absent from baseline, or appear to worsen from baseline during the study period

SECONDARY OUTCOMES:
Abstinence rate | 6 weeks
  It will be calculated by dividing the number of non-drinking days recorded during intervention by the total number of intervention days and multiplying the result by 100.
Average number of drinks consumed per day | 6 weeks
  Calculated as the total number of drinks during the intervention period divided by the total number of intervention days.
The number of drinking days | 6 weeks
  Calculated by counting the number of days on which a participant consumes alcohol during the intervention period.
The number of heavy drinking days | 6 weeks
  The number of heavy drinking days during the intervention period (having 3 or more drinks per day for males and 4 or more drinks per day for females.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong